CLINICAL TRIAL: NCT03111394
Title: A Pilot Study Evaluating the Feasibility of A Mobile Application to Collect Clinical, Magnetic Resonance Imaging Information and Genetic Data in Participants With Multiple Sclerosis
Brief Title: Study of myMS in Participants With a Diagnosis of Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Daniel Pelletier, Professor of Neurology; Vice Chair, Clinical Research, Department of Neurology; Division Chief, Neuro-Immunology and USC Multiple Sclerosis Center, University of Southern California
Other Study IDs: HS-16-00579
Record Dates: First submitted 2017-03-15; First posted 2017-04-12 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Multiple Sclerosis
Keywords: MS; 23andMe; MRI; Genome-wide association studies
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples are collected for DNA analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a pilot study looking at the feasibility of a mobile application (app) to collect data from active tasks (questionnaires, 6Mapp™, COGapp™, VISapp™), clinical magnetic resonance imaging information and conduct genome-wide association studies in subjects with multiple sclerosis. Participants will be self-referred to this study from different sources; patient advocacy groups, social media tools, clinicaltrials.gov, and flyers.

DETAILED DESCRIPTION:
This is a pilot study evaluating the feasibility of a mobile application "myMS™" to collect active clinical tasks (questionnaires, 6Mapp™, COGapp™, VISapp™), magnetic resonance imaging information and conduct genome-wide association studies in subjects with multiple sclerosis. Participants will be self-referred to this study from different sources; patient advocacy groups, social media tools, clinicaltrials.gov, and flyers.

Specific aims of this pilot study are:

1. To determine the feasibility and work flow in prospectively collecting surveys, clinical tasks, magnetic resonance imaging (MRI) information for up to 200 self-referred adult MS participants, using mobile app myMS™.
2. To determine the feasibility of using interface between myMS™ and 23andMe® DNA Kits and 23andme password protected mobile app platform (GSR Dashboard) in collecting one biological (saliva) sample and distributing the genetic result (using commercially available results only, distributed by 23andme®), for up to 200 self-referred adult MS participants. This aim is for testing the system interface only. 23andme® has their own independent consent form and IRB coverage for their commercial product.
3. To estimate the percentage of registered participants that will meet eligibility criteria for MS.
4. To estimate the percentage of participants that a) complete all clinical tasks; b) complete all surveys; c) provide genetic information; and d) provide MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* Males or females participants with access to an iPhone 5 and above.
* Participants willing to provide electronic consent.
* Age 18 and above.
* A diagnosis of MS (Polman, 2010), with dissemination in time and space. CIS participants will be included if they fulfil 3 of the 4 MRI criteria for dissemination in space as per Polman et al. 2010.
* EDSS of between 0 and 8.0

Exclusion Criteria:

* Under 18 years of age
* Participants who do not consent to participate.
* Participants participating in ongoing MS clinical trials with non-approved drugs.
* Any concurrent illness, disability or clinically significant abnormality (including laboratory tests) that may prevent the subject from safely completing the assessments required by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of Multiple Sclerosis.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Participants willing to provide genetic and MRI data via myMS | 12 months
  Proportion of participants with both genetic and MRI data available

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pelletier, M.D., Principal Investigator — Keck School of Medicine of USC, University of Southern California
Locations (1):
- Aimslab@Usc.Edu, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Participants will have the option to opt in or out for researchers to be able to share individual participant data (IPD) with researchers outside of USC.